CLINICAL TRIAL: NCT06056648
Title: Skin Images and Nomenclature for Diverse Populations (SkIN DP)
Brief Title: Addressing Inequity in Dermatology
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Dowager Countess Eleanor Peel Trust (Unknown)
Responsible Party: Principal Investigator, Elise Kleyn, Chief Investigator, University of Manchester
Other Study IDs: NHS001958
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dermatologic Disease
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are to understand the variation in dermatoses presenting in individuals from different ancestry backgrounds. This will be conducted at multiple NHS hospitals in England. The Investigators specifically aim to 1) assess features of dermatoses in individuals of different ancestry. 2) Understand the language used by patients describing their condition.

ELIGIBILITY:
Inclusion Criteria:

* Dermatologist diagnosed disease, with visible active dermatological disease

Exclusion Criteria:

* No dermatological disease, no active pathology identifiable, aged 18 and above but lacks capacity to consent.

Ages: 7 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dermatologist diagnosed dermatological condition with active disease and with clear morphology, of all ages and ancestries/ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assess features of dermatoses in individuals of different ancestry | Baseline
  Conducted through visual inspection of photographic images taken of the dermatological condition.
Asses the language used by patients when describing their skin condition | Baseline
  Content analysis and a framework analysis approach will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Chiedu Ufodiama, MBBS M.Sci, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided